CLINICAL TRIAL: NCT00159965
Title: Treatment for Psychogenic Nonepileptic Seizures: A Pilot, 12 Week, Prospective, Randomized, Placebo-controlled, Double-blind, Clinical Trial of Sertraline in the Treatment of Comorbid Psychiatric Disorders in NES
Brief Title: Treatments for Psychogenic Nonepileptic Seizures (NES)
Acronym: NES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, W. Curt LaFrance Jr., M.D., PI, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5K23NS045902-05 (NIH); 5K23NS045902 (NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Convulsion, Non-Epileptic; Conversion Disorder; Depression; Stress Disorders, Post-Traumatic
Keywords: nonepileptic seizure; pseudoseizure; conversion disorder; psychogenic; Depression; Anxiety; Abuse; post-traumatic stress disorder; sertraline; serotonin; randomized controlled trial
MeSH Terms: conditions — Seizures; Conversion Disorder; Depression; Stress Disorders, Post-Traumatic; Psychogenic Nonepileptic Seizures; Anxiety Disorders | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sertraline (Active Comparator): flexible dose sertraline, 25 to 200mg titration as tolerated, administered over 12 weeks with a two week untreated lead in period monitoring their baseline NES
  Interventions: Drug: sertraline
- placebo (Placebo Comparator): flexible dose placebo, administered over 12 weeks with a two week untreated lead in period monitoring their baseline NES
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sertraline — flexible dose sertraline
  Other Names: Zoloft
  Arms: sertraline
Drug: placebo — flexible dose placebo
  Arms: placebo

SUMMARY:
The investigators propose that treatment of the comorbid disorders (depression, anxiety, and impulsivity) with sertraline in patients with lone psychogenic nonepileptic seizures (NES), will result in a decreased number of NES. The purpose of this study is to provide pilot testing and data to inform the future randomized controlled trial based on the hypothesis.

DETAILED DESCRIPTION:
This is a pilot, prospective, single center, randomized, placebo-controlled, double-blind trial, that assesses the number of NES in patients treated with flexible dose sertraline (Zoloft). This study will provide outcomes data and the effect size necessary for a future R01, multi-center randomized control trial. Secondary objective variables include reduction in depression, anxiety, impulsivity scores, and improvement in psychosocial functioning.

After being diagnosed with NES by video electroencephalogram monitoring (vEEG), up to 50 participants will be enrolled and monitored during a two week lead in period for their baseline NES and psychosocial symptoms and functioning. At week 2, they will be blindly randomized to the treatment arm with flexible dose sertraline (25 to 200mg) or to the placebo control arm. The dose will be titrated over 4 weeks up to 200mg or to dose limited by side effects. The subjects will stay on their maximum fixed dose for the next 4 weeks. At week 10, the subjects may elect to remain on the sertraline or they can taper off the medication over the final two weeks of the treatment trial.

After the treatment trial, the subjects will have follow up phone calls at month 4, 8, and 12 after enrollment to assess seizure status, medication usage, and global functioning.

Upon enrollment, subjects will be evaluated with a structured psychiatric and neurological exam, and with bi-weekly, 30 to 60 minute appointments where they will complete symptom and function scales. They will keep a seizure diary prospectively, to evaluate their daily seizure activity. They will be given two weeks of the medication at each visit.

In the first phase of the study 12 patients were screened and 8 enrolled in an open label trial of flexible dose sertraline. In the second phase of the study, 38 patients enrolled in the pilot, randomized, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Video electroencephalogram (vEEG) confirmed diagnosis of NES
* Have at least one nonepileptic seizure per month
* Comorbid diagnosis of either depression, anxiety, or post traumatic stress disorder (PTSD)
* Able to complete self report symptom scales
* Not receiving optimized antidepressant medication

Exclusion Criteria:

* Equivocal electroencephalogram (EEG) findings
* Current suicidality, litigation, or self-mutilation
* Using monoamine oxidase inhibitors (MAOIs), pimozide, or sumatriptan
* Allergy/sensitivity to sertraline
* Current alcohol/drug dependence
* Serious medical illness requiring current hospitalization

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-12; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Curt LaFrance, Jr., MD, MPH, Principal Investigator — Rhode Island Hospital/Brown Medical School
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] LaFrance WC Jr, Devinsky O. The treatment of nonepileptic seizures: historical perspectives and future directions. Epilepsia. 2004;45 Suppl 2:15-21. doi: 10.1111/j.0013-9580.2004.452002.x. PMID 15186340
- [Background] LaFrance WC. How many patients with psychogenic nonepileptic seizures also have epilepsy? Neurology. 2002 Mar 26;58(6):990; author reply 990-1. doi: 10.1212/wnl.58.6.990. No abstract available. PMID 11914432
- [Background] LaFrance WC Jr, Alper K, Babcock D, Barry JJ, Benbadis S, Caplan R, Gates J, Jacobs M, Kanner A, Martin R, Rundhaugen L, Stewart R, Vert C; NES Treatment Workshop participants. Nonepileptic seizures treatment workshop summary. Epilepsy Behav. 2006 May;8(3):451-61. doi: 10.1016/j.yebeh.2006.02.004. Epub 2006 Mar 15. PMID 16540377
- [Background] LaFrance WC Jr, Barry JJ. Update on treatments of psychological nonepileptic seizures. Epilepsy Behav. 2005 Nov;7(3):364-74. doi: 10.1016/j.yebeh.2005.07.010. Epub 2005 Sep 16. PMID 16150653
- [Background] LaFrance WC Jr, Rusch MD, Machan JT. What is "treatment as usual" for nonepileptic seizures? Epilepsy Behav. 2008 Apr;12(3):388-94. doi: 10.1016/j.yebeh.2007.12.017. Epub 2008 Feb 20. PMID 18282812
- [Background] LaFrance WC Jr. Psychogenic nonepileptic seizures. Curr Opin Neurol. 2008 Apr;21(2):195-201. doi: 10.1097/WCO.0b013e3282f7008f. PMID 18317280
- [Background] LaFrance WC Jr, Devinsky O. Treatment of nonepileptic seizures. Epilepsy Behav. 2002 Oct;3(5 Suppl):19-23. doi: 10.1016/s1525-5069(02)00505-4. PMID 12609316
- [Background] LaFrance WC Jr, Benbadis SR. Avoiding the costs of unrecognized psychological nonepileptic seizures. Neurology. 2006 Jun 13;66(11):1620-1. doi: 10.1212/01.wnl.0000224953.94807.be. No abstract available. PMID 16769930
- [Result] LaFrance WC Jr, Blum AS, Miller IW, Ryan CE, Keitner GI. Methodological issues in conducting treatment trials for psychological nonepileptic seizures. J Neuropsychiatry Clin Neurosci. 2007 Fall;19(4):391-8. doi: 10.1176/jnp.2007.19.4.391. PMID 18070841
- [Result] LaFrance WC Jr, Syc S. Depression and symptoms affect quality of life in psychogenic nonepileptic seizures. Neurology. 2009 Aug 4;73(5):366-71. doi: 10.1212/WNL.0b013e3181b04c83. PMID 19652140
- [Result] LaFrance WC Jr, Keitner GI, Papandonatos GD, Blum AS, Machan JT, Ryan CE, Miller IW. Pilot pharmacologic randomized controlled trial for psychogenic nonepileptic seizures. Neurology. 2010 Sep 28;75(13):1166-73. doi: 10.1212/WNL.0b013e3181f4d5a9. Epub 2010 Aug 25. PMID 20739647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were referred to the Rhode Island Hospital (RIH) neuropsychiatry/behavioral neurology clinic between July 2002 and June 2008, after being diagnosed with psychogenic nonepileptic seizures (PNES). PNES diagnosis was established by capturing at least one of the patient's typical PNES on video electroencephalogram (vEEG).
Period: Overall Study
Arm/Group | Sertraline | Placebo
Started | 19 | 19
Completed | 12 | 14
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline | Placebo | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (13.9) | 34.4 (12.6) | 36.2 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Nonepileptic Seizures (NES)
Description: psychogenic nonepileptic seizure (NES) frequency, collected prospectively, using a daily seizure calendar; aggregated into biweekly intervals.
Time Frame: bi-weekly at baseline and weeks 2, 4, 6, 8, 10, 12
Measure: Median (Standard Deviation); unit: seizures
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
seizures
  Baseline (retrospective 2 weeks prior) | 5.0 (43.5) | 6.0 (12.1)
  Week 2 (prospectively collected from day 1-14) | 3.0 (37.7) | 6.0 (8.5)
  Week 4 | 2.0 (31.5) | 5.0 (10.6)
  Week 6 | 1.0 (31.5) | 3.0 (16.4)
  Week 8 | 1.0 (24.4) | 3.0 (17.4)
  Week 10 | 2.5 (30.7) | 7.0 (12.4)
  Week 12 | 0.0 (20.3) | 6.0 (14.0)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Between-group seizure change. The primary hypothesis of this pilot randomized control trial (RCT) was to assess the magnitude of seizure frequency reduction by treatment, comparing placbo to sertraline. The alternative hypothesis is that patients treated with sertraline will show a significant decrease in seizures from baseline to exit; Test type: Superiority or Other; p = 0.29, Overdispersed Poisson Regression; Risk Ratio, log = 0.673, 95% CI 2-sided [-0.051 to 1.396], Standard Error of Mean 0.369
Statistical Analysis 2: Comparison: Sertraline; Within-group seizure change. The hypothesis is that patients treated with sertraline will show a significant decrease in seizures from baseline to exit; Test type: Superiority or Other; p = 0.03, Overdispersed Poisson Regression; Risk Ratio, log = -0.598, 95% CI 2-sided [-1.139 to -0.073], Standard Error of Mean 0.276
Statistical Analysis 3: Comparison: Placebo; Within-group seizure change. The hypothesis is that patients treated with placebo will not show a significant decrease in seizures from baseline to exit; Test type: Superiority or Other; p = 0.78, Overdispersed Poisson Regression; Risk Ratio, log = 0.077, 95% CI 2-sided [-0.431 to 0.571], Standard Error of Mean 0.252

2. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: The BDI-II assesses depression severity from "0" (no Depression-related symptom) to "3" (severe) on each question. The highest possible score is "51", relating to the worst outcome.
Time Frame: bi-weekly at baseline and weeks 2, 4, 6, 8, 10, 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
Units on a scale
  Baseline | 16.7 (13.0) | 22.1 (13.9)
  Exit | 11.7 (11.5) | 17.0 (13.3)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

3. Secondary Outcome: Modified Hamilton Depression Scale (MHRS)
Description: The MHRS assesses the severity of Depression-related symptoms from "0" (not present) to "2", "3" or "4" (severe) on each question. The highest possible score is "72", relating to the worst outcome.
Time Frame: Baseline and weeks 2, 6, 10 (total time frame of 12 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
units on a scale
  Baseline | 17.8 (21.0) | 16.8 (8.8)
  Exit | 11.6 (9.0) | 13.3 (8.4)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

4. Secondary Outcome: Global Assessment of Functioning (GAF)
Description: This GAF rating scale ranges from 0 (worst) to 100 (best) and is used for evaluating the overall functioning of a subject during a specified time period on a continuum from psychological or psychiatric sickness to health.
Time Frame: Baseline and weeks 2, 6, 10 (total time frame of 12 weeks)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
Units on a scale
  Baseline | 53.3 (10.3) | 49.1 (7.1)
  Exit | 56.8 (11.0) | 52.0 (7.9)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

5. Secondary Outcome: Davidson Trauma Scale (DTS)
Description: The DTS is a 17-item self-report scale measuring each Diagnostic and Stastical Manual of Mental Disorders-4th Edition (DSM-IV) symptom of post-traumatic stress disorder (PTSD) on 5-point frequency (0-not at all to 4-everyday) and severity (0-not at all distressing to 4-extremely distressing) scales. The highest possible score is 136 and relates to the worst outcome.
Time Frame: Baseline and weeks 2, 6, 10 (total time frame of 12 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
units on a scale
  Baseline | 52.5 (31.6) | 48.1 (40.0)
  Exit | 40.3 (36.9) | 43.4 (40.0)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

6. Secondary Outcome: Barratt Impulsivity Scale (BIS)
Description: The BIS is a 30 item self-report measure that characterizes four aspects of impulsiveness, and ranges from "rarely/ never" to "almost always" with a score of "1" to "4" possible on each question, giving a maximum possible score of 120 and minimum possible score of 30. Selected questions are reversed scored. Higher scores relate to a worse outcome.
Time Frame: Baseline and weeks 2, 6, 10 (total time frame of 12 weeks)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
Units on a scale
  Baseline | 57.8 (16.5) | 72.6 (17.8)
  Exit | 64.9 (13.2) | 66.2 (15.9)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

7. Secondary Outcome: Dissociative Experiences Scale (DES)
Description: The DES is a 28 item self-report questionnaire designed to quantify dissociative experiences which identifies disturbances in memory, identity, cognition, derealization, depersonalization, absorption and imagination. A visual analogue scale is used ranging from 0% ("This never happens to you") to 100% ("This always happens to you"). The score is divided by 28 items to yield a range of 0 to 100%, with a higher score relating to a higher degree of dissociation.
Time Frame: Baseline and weeks 2, 6, 10 (total time frame of 12 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
units on a scale
  Baseline | 21.0 (19.7) | 17.4 (11.0)
  Exit | 8.5 (13.2) | 12.1 (12.2)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

8. Secondary Outcome: Symptom Checklist 90 (SCL-90)
Description: The SCL-90 is a 90 item self-report clinical rating scale oriented toward symptomatic behavior of outpatients, assessing from "0" (not at all bothered) to "4" (extremely bothered). The highest possible overall score is 360 and relates to a worse outcome.
Time Frame: Baseline and weeks 2, 6, 10 (total time frame of 12 weeks)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
Units on a scale
  Baseline | 84.9 (73.3) | 109.4 (70.9)
  Exit | 78.9 (67.2) | 91.4 (77.2)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

9. Secondary Outcome: Oxford Handicap Scale (OHS)
Description: The OHS is a brief clinician scored assessment of symptoms and lifestyle interference and the 6 grades of disability are based on the modified Rankin Scale, ranging from "0" (no symptoms) to "5" (severe handicap). A higher score relates to a worse outcome.
Time Frame: Baseline and weeks 2, 6, 10 (total time frame of 12 weeks)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
Units on a scale
  Baseline | 3.1 (0.8) | 3.4 (0.7)
  Exit | 2.3 (1.3) | 2.6 (1.2)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

10. Secondary Outcome: Clinical Global Impressions - Severity (CGI-S)
Description: The CGI-S is the first item of a two-item global rating scale, where each item is on a 7 point scale ranging from normal ("1") to among the most extremely ill patients ("7"). A higher score relates to a higher severity of illness.
Time Frame: Baseline and weeks 2, 6, 10 (total time frame of 12 weeks)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
Units on a scale
  Baseline | 4.9 (0.8) | 5.1 (0.6)
  Exit | 3.3 (1.6) | 3.9 (0.9)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

11. Secondary Outcome: Clinical Global Impressions - Improvement (CGI-I)
Description: The CGI-I is the second item of a two item global rating scale, where each item is on a 7 point scale ranging from very much improved ("1") to very much worse ("7"). A lower score represents a higher improvement.
Time Frame: Weeks 2, 6, 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
Units on a scale | 2.9 (1.4) | 3.5 (1.6)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

12. Secondary Outcome: Family Assessment Device (FAD)
Description: The FAD is a 60 item self-report questionnaire designed to assess the six dimensions of the McMaster Model of Family Functioning, as well as overall level of family functioning through the General Functioning Scale. Each question is scored on a "1" to "4" scale, with a higher mean score relating to a worse general functioning.
Time Frame: Baseline and weeks 2, 6, 10 (total time frame of 12 weeks)
Measure: Mean (Standard Deviation); unit: General Functioning Subscale Score
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
General Functioning Subscale Score
  Baseline | 2.0 (0.7) | 2.0 (0.5)
  Exit | 2.0 (0.6) | 2.2 (0.5)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

13. Secondary Outcome: Longitudinal Interval Follow-Up Evaluation Range of Impaired Functioning Tool (LIFE-RIFT)
Description: The LIFE-RIFT interview is a brief semi-structured interview, which measures functional impairment, targeting four domains: work, interpersonal relations, recreation and global satisfaction. Work, recreation and global satisfaction are rated on a "1" (very good/ no impairment) to "5" (very poor/ severe impairment) scale, and interpersonal relations is rated on a "1" (very good) to "7" (variable) scale. The highest score possible is 20 and relates to a more severe impairment. The lowest possible score is 3.
Time Frame: Baseline and weeks 2, 6, 10 (total time frame of 12 weeks)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
Units on a scale
  Baseline | 11.8 (3.6) | 13.9 (3.8)
  Exit | 11.8 (4.8) | 13.8 (3.3)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

14. Secondary Outcome: Quality of Life in Epilepsy-31 (QOLIE-31)
Description: This is a 31-item self-report scale used in the seizure population to evaluate Quality of Life. The lowest possible score is 0 and the highest possible score is 100, reflecting a better quality of life.
Time Frame: Baseline and weeks 2, 6, 10 (total time frame of 12 weeks)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 19 | 19
Units on a scale
  Baseline | 48.4 (20.7) | 38.2 (19.0)
  Exit | 56.7 (25.1) | 46.9 (24.0)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Sertraline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 1/19 | 4/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=19) | Placebo (N=19)
tiredness/ sleepiness (Nervous system disorders) | 1 (1) | 4 (4) — Adverse events profile and symptoms checklist

LIMITATIONS AND CAVEATS:
pilot sample size; drop-outs because of some patient's concern that they would receive the placebo, despite the equipoise that exists for NES treatment(s). Excluding patients who did not have vEEG may present a potential sampling bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No